CLINICAL TRIAL: NCT03799302
Title: Facilitating Sustainment Through Implementation Feedback: The SIC Coaching Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Responsible Party: Principal Investigator, Lisa Saldana, Principal Investigator, Oregon Social Learning Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R01DA044745 (NIH)
Record Dates: First submitted 2018-12-13; First posted 2019-01-10 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Evidence Based Practice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Consultation (No Intervention): Sites in this arm will receive the standard consultation from the TFCO or MDFT purveyors
- SIC Coaching Consultation (Experimental): In addition to the standard consultation from the TFCO or MDFT purveyors, sites in this arm will also receive feedback on how they are doing in terms of completing expected activities in their efforts to implement the designated EBP.
  Interventions: Behavioral: SIC Coaching

INTERVENTIONS:
Behavioral: SIC Coaching — Sites receiving consultation to implement either TFCO or MDFT will also receive consultation on their implementation fidelity as measured and tracked by the SIC.
  Arms: SIC Coaching Consultation

SUMMARY:
This study aims to test the impact of an empirically derived implementation strategy-under real-world conditions and across multiple child service systems-on successful adoption and sustainment of two evidence-based programs that address adolescent substance abuse: Treatment Foster Care Oregon (TFCO; formerly Multidimensional Treatment Foster Care) and Multidimensional Family Therapy (MDFT), both developed with funding from NIDA. Methods for this study utilize "technology-based approaches" for "implementing large-scale change." Leveraging previous data focused on developing and testing the 8-staged Stages of Implementation Completion (SIC) tool, a randomized evaluation of a SIC Coaching Strategy (SIC-CS) is proposed. Study activities include extending the SIC into the Sustainment Phase and testing the SIC-CS to support the adoption of new evidence-based programs.

ELIGIBILITY:
Inclusion Criteria:

* Senior leadership staff from teams that either currently are sustaining or who achieve 1-year sustainment post certification during the first year of the project

Exclusion Criteria:

* none

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Stages of Implementation Completion (SIC) | Baseline through month 60
  The SIC is an 8-stage observational assessment tool recording organizational site completion of implementation activities that map onto the three phases of implementation (Pre-Implementation, Implementation, Sustainability).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Saldana, PHD, Principal Investigator — Oregon Social Learning Center
Locations (1):
- Oregon Social Learning Center, Eugene, Oregon, United States